CLINICAL TRIAL: NCT03848260
Title: A Real-Time Magnetic Device Prototype for Management of Paralytic Lagophthalmos
Brief Title: A Real-Time Magnetic Device Prototype for Temporary Management of Paralytic Lagophthalmos
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Although six patients completed the test using device prototype before Dec 2019, but due to the large size and shape, we failed to well miniaturize and manufacture a resilient system that stands the test of time for the future trial.
Sponsor: E-DA Hospital (Other)
Collaborators: National Yang Ming Chiao Tung University (Other); The Industrial Technology Research Institute (Other); I-Shou University (Other)
Responsible Party: Principal Investigator, Lien, Ching-Feng, Deputy head of the Department of Otolaryngology-Head and Neck Surgery, E-Da Hospital, E-DA Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMRP33106N
Record Dates: First submitted 2019-02-13; First posted 2019-02-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Paralytic Lagophthalmos
Keywords: Lagophthalmos; Incomplete eye closure; Magnetic device; Blink restoration; Facial nerve palsy
MeSH Terms: conditions — Lagophthalmos; Bell Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Determine device feasibility (Experimental): by evaluating efficacy and safety of the device prototype. Test the device one time (duration: 60-120 mins/each time) and second time within 12 months.
  Intervention: using the magnetic device prototype
  Interventions: Device: Magnetic device prototype

INTERVENTIONS:
Device: Magnetic device prototype — The device prototype comprises a near-infrared light-emitting diode (SMT910, Epitex Inc, Kyoto, Japan) and receiver (PD15-22C TR8, Everlight Electronics Corporation, New Taipei City, Taiwan), a permanent electromagnetic actuator (JNP-12/12, Joint Magnetic Technology Corporation, Shenzhen, China), an iron sheet affixed to the paralytic upper eyelid, and a bio-signal acquisition module. The efficacy and safety of the device prototype was assessed using the device prototype.

SUMMARY:
To develop a real-time wearable device based on the principle of magnetic force for temporary management of lagophthalmos, and evaluate its efficacy and safety, including synchronous blinks and eye closure, blurred vision, foreign body sensation over cornea or eyeball, burning or hot sensation over facial skin, and erythema or pruritus over eyelid, by performing a human trial on patients with lagophthalmos.

DETAILED DESCRIPTION:
The wearable system includes a near-infrared (NIR) light-emitting diode (SMT910, Epitex Inc, Kyoto, Japan) and receiver (PD15-22C TR8, Everlight Electronics Corporation, New Taipei City, Taiwan), a permanent electromagnetic actuator (JNP-12/12, Joint Magnetic Technology Corporation, Shenzhen, China), an iron sheet affixed to the paralytic upper eyelid, and a bio-signal acquisition module together with a power supply unit providing a wired connection to the NIR sensor and permanent electromagnetic actuator. The palpebral gap was measured before and after the wearing of the device. The efficacy of the device prototype was assessed in terms of synchronous blinks and eye closure. Subjective sensation and complications were assessed by blurred vision, foreign body sensation over cornea or eyeball, burning or hot sensation over facial skin, and erythema or pruritus over eyelid. After the completion of the study procedure, eyelid skin condition was examined.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unilateral lagophthalmos; they are capable of understanding and complying with protocol requirements
* Aged 18 years old or older

Exclusion Criteria:

* Upper eyelid scar, contracture, fibrosis, and atrophy due to previous surgical intervention(s)
* Patients with psychiatric (or mental) disorders; they are unable to cooperate or follow the study procedure
* Children younger than 18 years of age

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in palpebral gap from the baseline. | 10 minutes after completion of the testing
  The investigators assess changes in distance between the upper and lower eyelid margins at the axis of the pupil (palpebral gap, millimeter) before and during the intervention by a ruler and/or a software.
Changes in visual acuity (blurred vision) from the baseline. | 10 minutes after completion of the testing
  Assess visual acuity by Snellen test before and after the intervention.
Discomfort of the eyeball and condition of the upper eyelid and facial skin based on a dichotomous Likert scale. | 10 minutes after completion of the testing
  The investigator assess discomfort of the eyeball, and examine erythema or swelling over upper eyelid and facial skin after the intervention. (The score 0 indicating no discomfort, score 1 indicating positive discomfort)
Changes in palpebral gap from the baseline. | 10 minutes after completion of the second testing within 12 months
  The investigators assess changes in distance between the upper and lower eyelid margins at the axis of the pupil (palpebral gap, millimeter) before and during the intervention by a ruler and/or a software.
Changes in visual acuity (blurred vision) from the baseline. | 10 minutes after completion of the second testing within 12 months
  Assess visual acuity by Snellen test before and after the intervention.
Discomfort of the eyeball and degree of the upper eyelid and facial skin based on a 3-point Likert scale. | 10 minutes after completion of the second testing within 12 months
  The investigator assess discomfort of the eyeball, and examine erythema or swelling over upper eyelid and facial skin after the intervention. The scale ranges from 1 to 3, with score 1 indicating no discomfort at all, score 2 moderate discomfort, and score 3 extremely discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Kun Tu, MD, Study Chair — E-Da Hospital, Kaohsiung, Taiwan
Locations (1):
- E-DA Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No